CLINICAL TRIAL: NCT00191529
Title: Optimization of Growth Hormone Treatment in Short Children Born Small for Gestational Age Based on a Growth Prediction Model-The OPTIMA Trial
Brief Title: Growth Hormone Treatment in Short Children Born Small for Gestational Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6581; B9R-EW-GDGB
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-06-15 (Estimated); Status verified 2007-06

CONDITIONS: Infant, Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

INTERVENTIONS:
Drug: somatropin

SUMMARY:
Comparison of 2 different doses of human growth hormone treatment on change in height after 1 and 2 years of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Born small for gestational age
* actual body height less than or equal -3 SDS
* chronological age greater than 3 years

Exclusion Criteria:

* Growth hormone deficiency
* any defined syndromal disease
* Diabetes mellitus

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2002-12; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The 2 different doses used are non-inferior to each other

SECONDARY OUTCOMES:
Safety profiles
Compare absolute height velocity

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne, Germany

REFERENCES:
- [Derived] Jung H, Land C, Nicolay C, De Schepper J, Blum WF, Schonau E. Growth response to an individualized versus fixed dose GH treatment in short children born small for gestational age: the OPTIMA study. Eur J Endocrinol. 2009 Feb;160(2):149-56. doi: 10.1530/EJE-08-0301. Epub 2008 Nov 27. PMID 19039085
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com